CLINICAL TRIAL: NCT07106151
Title: Outpatient Recovery From Acute Kidney Injury Requiring Dialysis - 2
Acronym: ORKID-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-44531; 5K23DK128605 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: AKI; AKI - Acute Kidney Injury; Dialysis Patients
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional AKI-D recovery information (Experimental)
  Interventions: Behavioral: Transmission of additional AKI-D recovery information
- No additional AKI-D recovery information (Active Comparator)
  Interventions: Other: No additional AKI-D recovery information

INTERVENTIONS:
Behavioral: Transmission of additional AKI-D recovery information — Measuring residual kidney function at the time of hospital discharge by timed urine collection (6-24 hours in duration), transmitting the results (urine volume, urea clearance, and creatinine clearance) to the accepting nephrologist and to the patient, along with information on recommended recovery monitoring frequency and criteria for consideration of a twice-weekly hemodialysis schedule.
  Arms: Additional AKI-D recovery information
Other: No additional AKI-D recovery information — The same timed urine collection will be collected at the time of hospital discharge as in the intervention arm, but in the control arm the results will not be transmitted to the accepting nephrologist or to the patient and no information on recommended recovery monitoring frequency and criteria for consideration of a twice-weekly hemodialysis schedule will be transmitted. Instead, the research team will call the accepting nephrologist to alert them that this is an AKI-D patient that is being followed by the research team for recovery for up to 60 days.
  Arms: No additional AKI-D recovery information

SUMMARY:
Providing additional information to patients with acute kidney injury who continue dialysis after hospital discharge and to the accepting kidney doctor (nephrologist) who manages their dialysis may be feasible and beneficial. This study will pilot measuring the patient's residual kidney function at the time of discharge and communicating that result to the accepting nephrologist and the patient, along with information on recommended recovery monitoring frequency and criteria for consideration of a twice-weekly hemodialysis schedule.

ELIGIBILITY:
Inclusion Criteria:

* AKI-D (not ESKD, as determined by the clinical inpatient nephrology team)
* Age ≥ 18 years
* Planned for continued dialysis outside the acute hospital setting (at outpatient dialysis unit/SNF/LTACH, not planned transfer to another short-stay acute care hospital).

Exclusion Criteria:

* Pregnant
* Prisoner
* Unable to consent and no surrogate decision maker available
* Clinical team declines to allow approach for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: The proportion of patients who complete the timed urine collection within seven days before discharge and are able to have the results successfully transmitted to the accepting nephrologist and patient. | Baseline

SECONDARY OUTCOMES:
Recruitment rate: Number of patients enrolled per month | Total study duration, anticipated 2 years
Screening-to-recruitment ratio: Number of patients who meet inclusion criteria divided by the number of patients enrolled. | Total study duration, anticipated 2 years
Number of post-discharge urine collections completed | Study day 60
Proportion prescribed a <3x/wk hemodialysis schedule at any time within 60 days of hospital discharge | Study day 60
Proportion who recover from needing dialysis | Study day 60
Proportion who trial a <3x/wk hemodialysis schedule but subsequently need to be increased to >= 3x/wk during the 60-day follow-up. | Study day 60
Incidence of adverse events | Study day 60

CONTACTS AND LOCATIONS:
Overall Officials: Ian E McCoy, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No